CLINICAL TRIAL: NCT00940667
Title: A Phase III, 8-week, Multicenter, Randomized, Double-blind Study to Compare the Efficacy and Safety of Amlodipine 5mg+Losartan 50mg Versus Amlodipine 10mg in Patients With Essential Hypertension Not Controlled on Amlodipine Monotherapy
Brief Title: Efficacy/Safety of Amlodipine Plus Losartan Versus Amlodipine in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALOS-301
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: Amlodipine; Losartan; hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amlodipine/losartan 5/50mg (Experimental)
  Interventions: Drug: Amlodipine plus Losartan
- amlodipine 5mg (Active Comparator)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine plus Losartan — amlodipine/losartan 5/50mg q.d.
  Other Names: Amosartan
  Arms: amlodipine/losartan 5/50mg
Drug: Amlodipine — amlodipine 5mg q.d.
  Other Names: Amodpine
  Arms: amlodipine 5mg

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety of amlodipine plus losartan and amlodipine alone in patients with essential hypertension inadequately controlled on amlodipine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Essential hypertensive patients whose blood pressure is not controlled before the study (sit DBP ≥ 90 mmHg for drug-treated patient, sit DBP ≥ 95 mmHg for drug-naïve patient)
* Non-responder to 4 weeks treatment of amlodipine 5 mg monotherapy (sit DBP ≥ 90mmHg)

Exclusion Criteria:

* mean sit SBP ≥ 200 mmHg or mean sit DBP ≥ 120 mmHg at screening
* mean sit SBP ≥ 180 mmHg or mean sit DBP ≥ 120 mmHg after 4 weeks of amlodipine 5 mg treatment
* has a history of hypersensitivity to dihydropyridines or angiotensin II receptor blockers
* Secondary hypertensive patient or suspected to be
* Uncontrolled diabetes mellitus patients
* Severe heart disease or severe neurovascular disease
* Known as severe or malignant retinopathy
* Patients showed clinically significant hematological finding, patients with renal diseases (serum creatinine), patients with hepatic disease (ALT or AST)
* History of malignancy tumor
* History of autoimmune disease
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, has an intention on pregnancy
* Considered by investigator as not appropriate to participate in the clinical study with othe reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure | Week 8

SECONDARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure | Week 4
Change from baseline in mean sitting systolic blood pressure | Week 4, 8
Responder rate | Week 4, 8

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yun Cho, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- 13 sites in Korea, Seoul, Busan, Etc., South Korea

REFERENCES:
- [Derived] Kang SM, Youn JC, Chae SC, Park CG, Yang JY, Kim MH, Hong TJ, Kim CH, Kim JJ, Shin DG, Jeong JW, Yoon JH, Park SH, Kwon J, Cho SY. Comparative efficacy and safety profile of amlodipine 5 mg/losartan 50 mg fixed-dose combination and amlodipine 10 mg monotherapy in hypertensive patients who respond poorly to amlodipine 5 mg monotherapy: an 8-week, multicenter, randomized, double-blind phase III noninferiority study. Clin Ther. 2011 Dec;33(12):1953-63. doi: 10.1016/j.clinthera.2011.11.007. Epub 2011 Dec 2. PMID 22136978